CLINICAL TRIAL: NCT07022977
Title: A Randomized, Double-blind, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MET233 in Otherwise Healthy Adult Participants With Obesity or Overweight
Brief Title: A Study of MET233 in Individuals With Obesity or Overweight
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Metsera, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MET233-24-101
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Part A (40 participants), Part B (40 participants), Part C (40 participants)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- (Part A) MET233 (Experimental): Participants will receive a single dose of MET233 at up to 5 dose levels
  Interventions: Biological: MET233
- (Part A) Placebo (Placebo Comparator): Participants will receive a single dose of placebo
  Interventions: Biological: Placebo
- (Part B) MET233 (Experimental): Participants will receive five weekly doses of MET233 at up to 4 dose levels
  Interventions: Biological: MET233
- (Part B) Placebo (Placebo Comparator): Participants will receive five weekly doses of placebo
  Interventions: Biological: Placebo
- (Part C) MET233 (Experimental): Participants will receive twelve weekly doses of MET233 at up to 4 dose levels, followed by a 13th potential monthly dose
  Interventions: Biological: MET233
- (Part C) Placebo (Placebo Comparator): Participants will receive twelve weekly doses of placebo, followed by a 13th potential monthly dose
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MET233 — For subcutaneous administration
  Arms: (Part A) MET233; (Part B) MET233; (Part C) MET233
Biological: Placebo — Sterile 0.9% (w/v) saline for subcutaneous administration
  Arms: (Part A) Placebo; (Part B) Placebo; (Part C) Placebo

SUMMARY:
The goal of this clinical trial is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of once-weekly subcutaneous injections of MET233 in otherwise healthy adults with overweight or obesity.

The trial will be conducted in three parts. Part A consists of single ascending dose (SAD) cohorts of MET233 or placebo. Part B consists of multiple ascending dose (MAD) cohorts, with participants treated with five once-weekly doses of MET233 or placebo. In Part C, participants will receive once-weekly doses of MET233 or placebo for 12 weeks, followed by a single higher, potential monthly dose.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind study designed to investigate the safety, tolerability, PK and pharmacodynamic (PD) of single and multiple ascending subcutaneous (SC) doses of MET233 in otherwise healthy adult participants with obesity or overweight (body mass index [BMI] 27.0 kg/m2 to 38.0 kg/m2, inclusive).

In Part A, approximately 40 participants will receive a single dose of MET233 at up to 5 dose levels. In Part B, approximately 40 participants will receive five weekly doses of MET233 at up to 4 dose levels. In Part C, up to 4 cohorts of 10 participants each will receive 12 weekly doses. These doses may include titration. For all cohorts in Part C, the 13th dose of MET233 administered on Day 85 may be a monthly-equivalent dose to allow evaluation of a potential to switch to a monthly dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 to ≤70 years) male and female participants with obesity or overweight (BMI 27.0 kg/m2 to 38.0 kg/m2, inclusive) but otherwise healthy.

Exclusion Criteria:

* Female who is lactating or who is pregnant according to the pregnancy test at the Screening visit or prior to the first study drug administration
* Seated blood pressure higher than 160/95 mmHg at the Screening visit
* Elevated resting pulse greater than 100 beats per minute at Screening visit
* Presence of clinically significant ECG abnormalities
* Diagnosis of diabetes (type 1 or type 2)
* Participation in a weight loss program with or without pharmacotherapy during the 3 months prior to study administration
* Obesity induced by endocrinologic disorders (e.g., Cushing's syndrome) or diagnosed monogenetic or syndromic forms of obesity (e.g., Melanocortin 4 Receptor deficiency or Prader-Willi Syndrome).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events | Part A - Baseline (Day 0) to Day 89 Part B - Baseline (Day 0) to Day 113 Part C - Baseline (Day 0) to Day 162

SECONDARY OUTCOMES:
Area under the concentration versus time curve during the dosing interval (AUC(0-τ)) | Part A: Baseline (Day 0) to Day 85 Part B: Baseline (Day 0) to Day 113 Part C: Baseline (Day 0) to Day 162
Maximum observed concentration (Cmax) | Part A: Baseline (Day 0) to Day 85 Part B: Baseline (Day 0) to Day 113 Part C: Baseline (Day 0) to Day 162
Time to maximum observed concentration (Tmax) | Part A: Baseline (Day 0) to Day 85 Part B: Baseline (Day 0) to Day 113 Part C: Baseline (Day 0) to Day 162
Elimination half-life (t1/2) | Part A: Baseline (Day 0) to Day 85 Part B: Baseline (Day 0) to Day 113 Part C: Baseline (Day 0) to Day 162
Percent change from baseline in body weight at the protocol-specified weekly post-baseline measurements | Part A: Baseline (Day 0) to Day 85 Part B: Baseline (Day 0) to Day 113 Part C: Baseline (Day 0) to Day 162

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- MET233 Research Site 001, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Undecided